CLINICAL TRIAL: NCT05497453
Title: Phase 1/2 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of OTX-2002 As a Single Agent and in Combination with Standard of Care in Patients with Hepatocellular Carcinoma and Other Solid Tumor Types Known for Association with the MYC Oncogene
Brief Title: A Phase 1/2 Study to Evaluate OTX-2002 in Patients with Hepatocellular Carcinoma and Other Solid Tumor Types Known for Association with the MYC Oncogene
Acronym: MYCHELANGELO I
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate after monotherapy dose escalation.
Sponsor: Omega Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTX-2002-101
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma; Solid Tumor; Hepatocellular Carcinoma Non-resectable; Hepatocellular Carcinoma Recurrent; Hepatocellular Cancer; Liver Cancer; Liver, Cancer Of, Non-Resectable
Keywords: MYC; C-MYC; MYC Amplification; MYC Overexpression; MRNA; Epigenetics
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Part 1 OTX-2002 monotherapy dose escalation and expansion in participants with hepatocellular carcinoma (HCC) and other solid tumors
  During the monotherapy dose escalation phase, participants will be enrolled in sequential cohorts of increasing doses of OTX-2002.
  Part 2 of the study is a safety run-in and expansion study of OTX-2002 participants with HCC will be administered OTX-2002 in combination with tyrosine kinase inhibitor One (Part 2A), Tyrosine Kinase Inhibitor Two (Part 2B), or Checkpoint Inhibitor (Part 2C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- OTX-2002 (Experimental): Monotherapy: OTX-2002 (Cycle length = 4 weeks) OTX-2002 will be administered as an IV infusion over 80-120 minutes every 2 weeks
  Interventions: Drug: OTX-2002
- OTX-2002 + Tyrosine Kinase Inhibitor One (Experimental): OTX-2002 + Tyrosine Kinase Inhibitor One: (Cycle length = 4 weeks) OTX-2002 will be administered as an IV infusion over 80-120 minutes every 2 weeks.
  Tyrosine Kinase Inhibitor One will be standard per the respective fixed local approved dose
  Interventions: Drug: OTX-2002; Drug: Tyrosine kinase inhibitor One
- OTX-2002 + Tyrosine Kinase Inhibitor Two (Experimental): OTX-2002 + Tyrosine Kinase Inhibitor Two : (Cycle length = 4 weeks) OTX-2002 will be administered as an IV infusion over 80-120 minutes every 2 weeks.
  Tyrosine Kinase Inhibitor Two will be standard per the respective fixed local approved dose
  Interventions: Drug: OTX-2002; Drug: Tyrosine kinase inhibitor Two
- OTX-2002 + Checkpoint Inhibitor (Experimental): OTX-2002 + Immune Checkpoint Blockade: (Cycle length = 6 weeks) OTX-2002 will be administered as an IV infusion over 80-120 minutes every 2 weeks.
  Checkpoint Inhibitor will be standard per the respective fixed local approved dose
  Interventions: Drug: OTX-2002; Drug: Checkpoint Inhibitor, Immune

INTERVENTIONS:
Drug: OTX-2002 — OTX-2002 is a lipid nanoparticle (LNP) that contains a biscistronic mRNA that codes for 2 independent epigenomic controllers.
Drug: Tyrosine kinase inhibitor One — Tyrosine Kinase Inhibitor
  Arms: OTX-2002 + Tyrosine Kinase Inhibitor One
Drug: Tyrosine kinase inhibitor Two — tyrosine kinase inhibitor
  Arms: OTX-2002 + Tyrosine Kinase Inhibitor Two
Drug: Checkpoint Inhibitor, Immune — monoclonal antibody that binds to PD-1 or PD-L1
  Arms: OTX-2002 + Checkpoint Inhibitor

SUMMARY:
This is a Phase 1/2 open-label study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of OTX-2002 as a single agent and in combination with standard of care in patients with hepatocellular carcinoma (HCC) and other solid tumor types known for association with the MYC oncogene.

The study consists of Part 1 (OTX-2002 monotherapy) and Part 2 (OTX-2002 combined with standard of care in hepatocellular carcinoma). Part 1 consists of escalation and expansion, and Part 2 consists of safety run-in and expansion. The objective of Part 1 escalation and Part 2 safety run-in will be safety and tolerability, while anti-tumor activity will be evaluated as the primary endpoint in Part 1 and Part 2 expansion.

DETAILED DESCRIPTION:
This is a Phase 1/2 open-label study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of OTX-2002 as a single agent and in combination with standard of care in patients with hepatocellular carcinoma (HCC) and other solid tumor types known for association with the MYC oncogene. The study consists of Part 1 (OTX-2002 monotherapy) and Part 2 (OTX-2002 combined with standard of care in hepatocellular carcinoma).

In Part 1, during dose escalation, participants with HCC and other solid tumors that progressed on, relapsed after, are refractory to, or are intolerant of standard of care for which no treatment options are available will be administered an intravenous infusion of OTX-2002 as a single agent. The escalation will be conducted using a 3+3 design, with the primary endpoint of dose limiting toxicity (DLT), maximum tolerated dose (MTD), and incidence of treatment emergent adverse events (TEAEs). In Part 1 expansion, 15-25 participants with BCLC stage B or C, Child-Pugh Class A HCC who have received at least 1 prior line of systemic anticancer treatment, and without available subsequent standard of care, will receive OTX-2002 at the recommended dose for expansion (RDE) for monotherapy. The primary endpoint of Part 1 expansion will be overall response rate (ORR) and duration of response (DoR).

In Part 2, during safety run-in, participants with BCLC stage B or C, Child-Pugh Class A HCC who have received at least 1 prior line of systemic anticancer treatment, and without available subsequent standard of care, will receive OTX-2002 at the selected dose in combination with standard of care therapies at the local approved dose. The primary endpoint of Part 2 safety run-in will be DLT, MTD, and incidence of TEAE. Once the combination therapies have been determined to be tolerable in the safety run-in, 15-25 HCC participants will be enrolled in Part 2 expansion for each of the combination therapies. The primary endpoint of Part 2 expansion will be ORR and DoR.

ELIGIBILITY:
Key inclusion

* Participants with metastatic, advanced (non-resectable), or recurrent solid tumor who progressed on, relapsed after, are refractory to, or intolerant of standard of care (only applicable to Part 1 escalation)
* Participants with BCLC Stage B (intermediate stage) or C (advanced stage), Child-Pugh A hepatocellular carcinoma who is not amenable to locoregional therapy, refractory to locoregional therapy or not amenable to curative treatment approach
* Adult participants age ≥ 18 years at the time of signing informed consent
* Participant must have progressed on, have relapsed after, be refractory to, or be intolerant of at least 1 prior systemic therapy, and without available subsequent standard of care
* Participants with chronic hepatitis B must have received antiviral therapy for hepatitis B virus (HBV) for at least 12 weeks and HBV viral load must be < 500 IU/mL prior to first dose of study drug.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Key exclusion

* Mixed histology cholangiocarcinoma and HCC, or fibrolamellar variant HCC
* Hepatocellular carcinoma with ≥ 50% liver occupation
* Clear invasion into the bile duct
* Portal vein invasion with Vp4
* Active/untreated CNS metastases or carcinomatous meningitis
* History of ascites requiring paracentesis within the past 3 months
* Esophageal or gastric variceal bleeding in the past 3 months
* History of hepatic encephalopathy in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Determine Dose limiting toxicities (DLT)and maximum tolerated dose ( MTD) (Part 1 escalation and Part 2 safety run-in) | 28 days/4 weeks from the first dose of OTX-2002
  The frequency of DLTs will be tabulated by dose for participants in the dose escalation phase, and information about all DLTs will be listed by dose.
Incidence of TEAEs including all AEs,Grade 3-5 AEs, drug-related AEs, and SAEs (Part 1 escalation and Part 2 safety run-in) | 30 days after the last dose of study drug
  The incidence of TEAEs, SAEs, and TEAEs leading to study drug discontinuation will be summarized for all patients.
Overall response rate (ORR)(for Part 1 and Part 2 expansion) | through treatment completion, up to two years
  ORR (proportion of participants who achieve CR or PR), DCR (proportion of participants who achieve CR, PR, or SD)per mRECIST (for HCC) and RECIST 1.1(for solid tumors), during Parts 1, 2A, 2B,and 2C
  •ORR (proportion of participants who achieve CR or PR), DCR (proportion of participants who achieve CR, PR, or SD)per irRECIST during Part 2C
Duration of Response (DOR) (for Part 1 and Part 2 expansion) | through treatment completion, up to two years
  Duration of Complete Response and Partial Response

CONTACTS AND LOCATIONS:
Overall Officials: Yan Moore, MD, Study Director — Omega Therapeutics
Locations (15):
- United States (6):
  - City of Hope, Duarte, California
  - University of Florida Health Cancer Center, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Stephenson Cancer Center at Oklahoma University, Oklahoma City, Oklahoma
  - Fred Hutch / University of Washington, Seattle, Washington
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Singapore (2):
  - National Cancer Center Singapore, Singapore
  - National University Hospital, Singapore
- South Korea (3):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided